CLINICAL TRIAL: NCT07047287
Title: Global Postural Reeducation Versus Pilates in Patients With Non-specific Low Back Pain
Acronym: LBP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, ibrahim mostafa mohamed, principle investigator : ibrahim mostafa mohamed, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005702
Record Dates: First submitted 2025-06-24; First posted 2025-07-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Low Back Pain
Keywords: global postural reeducation; pilates; low back pain
MeSH Terms: conditions — Low Back Pain | interventions — Exercise Movement Techniques

STUDY DESIGN:
Intervention Model Description: global postural reeducation and pilates
Who Masked: Outcomes Assessor
Masking Description: opaque sealed envelope
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- global postural reeducation exercise (Experimental): Twenty patients suffer from nonspecific low back pain and will be received Global postural reeducation exercise and conventional physiotherapy treatment two times a week for six weeks
  Interventions: Other: global postural reeducation exercise; Other: conventional therapy
- pilates exercises (Experimental): Twenty patients suffer from nonspecific low back pain and will receive Pilates exercise and conventional physiotherapy treatment two times a week for six weeks
  Interventions: Other: pilates exercises; Other: conventional therapy
- conventional therapy (Active Comparator): Twenty patients suffer from nonspecific low back pain and will receive conventional physiotherapy treatment two times a week for six weeks.
  Interventions: Other: conventional therapy

INTERVENTIONS:
Other: global postural reeducation exercise — The global postural reeducation exercise involves a sequence of active, moderate postures as well as exercises that are designed to realign joints, stretch shortened muscles, in addition, strengthen the contraction of the antagonist's muscles to prevent postural asymmetry. There are eight different therapeutic postures in the GPR approach that should be held for 15 to 20 min while lying, sitting, or standing. Only two or three postures have been proposed to encourage treatment standardization+ conventional therapy
  Arms: global postural reeducation exercise
Other: pilates exercises — the patients will receive pilates in the form of single leg stretch + Pelvic press + Swimming + Opposite arm and leg reach + Side to side), 3 sets of 10 repetitions
  Arms: pilates exercises
Other: conventional therapy — the patients will receive conventional physiotherapy treatment which consists of routine physical therapy eg. (Back, hamstring, calf and hip flexors stretches, Abdominal curl up exercises etc along with ultrasound and Transcutaneous electrical nerve stimulation (TENS).

SUMMARY:
to compare between Global Postural Reeducation and Pilates mat on pelvic angles, pain intensity, hip flexibility and Functional disability in patients with chronic non-specific low back pain

DETAILED DESCRIPTION:
Chronic low back pain is a common health problem in many developed and developing countries. Individuals suffering from chronic low back pain experience major physical, social, mental, and occupational disruptions. It is not only one of the leading causes of pain but also of a costly burden on the health care budget as chronic low back pain leads to a frequent demand for medical services. The majority of patients (up to 90%) are categorized as having nonspecific low back pain.Global postural reeducation (GPR) is a conservative treatment that we can consider as a global postural exercise method, and widely used in physical therapy clinical practice in many countries. Pilates is a concept of body and mind exercise and a system of repetitive exercises including whole-body movements, breathing, centering, rhythm, and concentration. Pilates is a mindful approach exercise that promote strength, stability and is used for health enhancement and in several diseases.

ELIGIBILITY:
Inclusion Criteria:

* 18-50 years old, Low back pain for more than 3 months (pain felt between T12 and the gluteal fold).
* Patients willing and able to participate in an exercise program safely and without cognitive impairments that would limit their participation.
* BMI index smaller than 30 kg/m2
* Both male and female gender were included in the study.
* Nonspecific, non-radicular (axial) chronic LBP diagnosis (LBP for at least three months).
* Visual Analog Scale (VAS) score of 3 or higher

Exclusion Criteria:

* History of back surgery
* Rheumatologic disorders,
* Spine infections
* Spine exercise training in the 3 months before the onset of the study.
* Under psychiatric care.
* Neurological conditions that would interfere with the assessments, such as major sensory changes, and level of consciousness/ understanding
* Advanced joint disease.
* History of severe physical and nervous system diseases
* Unable to cooperate with the study protocols.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-30 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
pain intensity | up to six weeks
  VAS is employed as a quantitative tool to assess the subjective intensity of pain experienced by an individual. The VAS is a reliable and valid method for assessing low back pain clinically. It consists of a single handwritten mark down the length of a 10-cm line, with "no pain" at one end of the scale (0 cm) and "worst pain" at the other (10 cm)

SECONDARY OUTCOMES:
disability | up to six weeks
  The Arabic version of the Oswestry Disability Index (ODI) has been applied to evaluate the disability brought reliability. The questionnaire was filled out by the patient in about 5 min, and the doctor scored it in around 1 min. Each component is given a score between 0 and 5, with 5 being the most severe disability. The index is determined through the division of the total score by the range of scores, and then its numerical representation as a percentage is derived by multiplying the result by 100. As a result, the denominator drops by 5 for each query that is unanswered
anterior pelvic tilt | up to six weeks
  Using the iHandy Level app on a smartphone will be used to assess anterior pelvic tilt. The anterior and posterior iliac spines were felt. The iHandy's angle was set to 0 while the patient was lying prone, and a semi-permanent pen was used to mark the skin at levels L5-S1.The patient was lying in a long sitting position with his or her feet flat against a wall. The examiner instructed the patient to move their ischial tuberosities into a more posterior position and to raise their chest towards the wall. Try to stay at the same height while you move forward from the hips. Proceed as far as you are able to. Stop when you feel you can no longer go or when your knees start to lift under your hands. Instead of bouncing, hold as tightly as you can. There were only 10 s in this pose.
lumbar lordosis | up to six weeks
  flexible ruler will be used to assess lumbar lordosis. To get an accurate reading of lumbar lordosis, a flexible ruler is employed. The flexible ruler demonstrates high reliability and validity as a portable and non-invasive tool for measuring lumbar lordosis. Specifically, the validity of lumbar lordosis measures obtained using the flexible ruler, when compared to those obtained using X-ray imaging, is reported to be 0.91. An angel's theta can be calculated using the formula [theta]=4×[arctan(2H/L)], where theta stands for the magnitude of the lordotic curve. The lumbar lordotic angle typically ranges from 6.50 to 17.80°.
hip flexor flexibility | up to six weeks
  hip flexor flexibility will be used to assess hip flexor flexibility. The modified Thomas test has been used to evaluate hip flexor flexibility. The patient was lying on their back during this test, and their thigh was hanging over the side of the examination table. The patient firmly held the thigh of the unexamined limb and brought it closer to their chest. The pelvis was rotated posteriorly, and the lumbar spine was flat on the plinth.
  Using a goniometer to measure the angle of hip flexion, the length of the iliopsoas muscle was determined. The femur's greater trochanter and fulcrum were in line. Using the pelvis as a reference point, the measurement was performed by positioning the goniometer's fixed arm along the lateral midline of the abdomen and its moving arm along the lateral midline of the femur.